CLINICAL TRIAL: NCT04855448
Title: Accelerated Learning Curve in Low Anterior Resection for Rectal Resection, a New Surgical Robot Micro Hand S Versus da Vinci, Can be Attained Simultaneously: a Single Center Experience
Brief Title: Evaluation of the Learning Curve in Low Anterior Resection for Rectal Resection With the Two Surgical Robots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XY3-DSRCS1507A04
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon A (Experimental): This group is consisted of 56 cases performed using the Micro Hand S robot and da Vinci robot by one single surgeon in low anterior resection for rectal cancer
  Interventions: Device: Micro Hand S robot and da Vinci robot
- Surgeon B (Active Comparator): This group is consisted of 56 cases performed using the da Vinci robot by one single surgeon in low anterior resection for rectal cancer
  Interventions: Device: da Vinci robot

INTERVENTIONS:
Device: Micro Hand S robot and da Vinci robot — The surgeries are performed with the Micro Hand S robot and da Vinci robot
  Arms: Surgeon A
Device: da Vinci robot — The surgeries are performed with the da Vinci robot
  Arms: Surgeon B

SUMMARY:
Central South University in collaboration with Tianjin University developed the first domestically produced Chinese minimally invasive surgical (MIS) robot system which named "Micro Hand S" in 2013. This new MIS robot had been authorized to enter the clinical trial stage by the Ethics Committee of the Third Xiangya Hospital at Central South University. The Micro Hand S robot is safe and feasible in the preliminary study. However, the learning curve in low anterior resection for rectal resection with the Micro Hand S robot are unclear and whether the two surgical robots (Micro Hand S and da Vinci) shared a similar learning curve and the two robot can be trained simultaneously. Therefore, the investigators conduct this retrospective study to focus on this concern.

DETAILED DESCRIPTION:
The Micro Hand S robor has been appiled in low anterior resection for rectal cancer. The safey and feasibility has been evaluated. However, the learning curve of this procedure is unclear. Specially,whether the two surgical robots (Micro Hand S and da Vinci) shared a similar learning curve and the two robot can be trained simultaneously are unclear.Therefore, this srudy is conducted to evaluate the learning curve of the two robots in low anterior resection.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed rectal cancer; ASA score ≤ 3

Exclusion Criteria:

* palliative resections, combined resections, distant metastasis, a previous history of abdominal/or pelvic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
learning curve of console time | up to 1 week after operation
  It was defined the cumulative sum plot of the consloe time in the chronological order.
learning curve of docking time | up to 1 week after operation
  It was defined the cumulative sum plot of the docking time in the chronological order.
learning curve of surgicla failure | up to 1 week after operation
  It was defined the cumulative sum plot of the docking time in the chronological order.

SECONDARY OUTCOMES:
Type of surgical procedure | up to 1 week after operation
  It was defined as what type of procedure was pferformed, for example, low anterior, abdominal perineal resection
Operative time (min) | up to 1 week after operation
  It was defined as the duration from skin incision to skin closure
Console time (min) | up to 1 week after operation
  The console time was defined the fime that the surgeon performed the surgeon console.
Docking time (min) | up to 1 week after operation
  The docking time was the time from moving robotic instruments in the surgical field to setting robotic arms into the port sites
Conversion | up to 1 week after operation
  Conversion was defined as any change in strategy to open surgery
Bloos loss (ml) | up to 1 week after operation
  It was defined as the amount of blood in the whole surgical time
Hospital stay (day) | up to 1 month after operation
  It was defined as the length of hospital stay
Protective ileostomy | up to 1 month after operation
  It was defined as ileostomy which diverted the feces to to ensure anastomotic healing
Retrieved lymph node | up to 1 month after operation
  It was defined as the number of all the lymph nodes for each patient
Surgical failure | up to 1 month after operation
  Surgical failure was defined as the presence of one or more of the following four parameters: conversion, the positive surgical margins, severe postoperative complications, the number of harvested lymph nodes less than 12
pTNM stage | up to 1 month after operation
  It was defined as the pathological stage of the tumor according the TNM classification
Tumor size (cm) | up to 1 month after operation
  It was defined as the longitudinal diameter of the tumor
Length of distal ressction margin (cm) | up to 1 month after operation
  It was defined as the distance betwen the distal resection margin and the low margin of the tumor
Status of the surgical margin | up to 1 month after operation
  It was defined as whether the distal and circumferential resection margins was involved the tumor cell under microscope
Quality of specimen | up to 1 month after operation
  The quality of the speciman was graded according to the protocol proposed by Quirke
Postoperative complication | up to 1 month after operation
  It was defined as the adverse events after operation and the complications were classfied according to the Clavien-Dindo (C-D) classification
Local recurrence | at least 1 years after operation
  It was defined as the tumor was again found in the pelvic cavity
Disease free survival | at least 1 years after operation
  It was defined as the duration between the operation and date of the tumor recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No